CLINICAL TRIAL: NCT01991678
Title: An Open-Label, Parallel-Group, Multicenter, Phase 1 Study to Investigate the Pharmacokinetics of NKTR-102 for Injection (Etirinotecan Pegol) in Patients With Advanced or Metastatic Solid Tumors and Hepatic Impairment
Brief Title: A Study in Cancer Patients With Hepatic Impairment to Evaluate the Pharmacokinetics and Safety of NKTR-102 (Etirinotecan Pegol)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nektar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-102-13
Record Dates: First submitted 2013-10-29; First posted 2013-11-25 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Advanced or Metastatic Solid Tumors in Patients With Hepatic Impairment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- normal hepatic function (Experimental): 12 Patients will receive a 90-minute IV infusion
  Interventions: Drug: 145 mg/m2 NKTR 102
- mild hepatic dysfunction (Experimental): 6 Patients will receive a 90-minute IV infusion
  Interventions: Drug: 120 mg/m2 NKTR 102
- severe hepatic dysfunction (Experimental): 6 Patients will receive a 90-minute IV infusion
  Interventions: Drug: 50 mg/m2 NKTR 102

INTERVENTIONS:
Drug: 145 mg/m2 NKTR 102
  Arms: normal hepatic function
Drug: 120 mg/m2 NKTR 102
  Arms: mild hepatic dysfunction
Drug: 50 mg/m2 NKTR 102
  Arms: severe hepatic dysfunction

SUMMARY:
The purpose of this study is to investigate the PK and safety of NKTR-102 in patients with mild, moderate, or severe hepatic impairment.

DETAILED DESCRIPTION:
Safety and PK data from patients with mild, moderate, or severe hepatic impairment will be compared with a control group consisting of patients with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or progressive advanced solid tumor malignancies
* Measurable or non-measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Life expectancy greater than 3 months
* Resolution of all acute toxic effects of prior chemotherapy, and other cancer treatments
* Adequate bone morrow and kidney function
* No signs of decompensated liver cirrhosis or ascites requiring therapeutic paracentesis
* Agree to use adequate contraception

Exclusion Criteria:

* Previous chemotherapy, immunotherapy, chemo-embolization, targeted therapy or investigational agent for malignancy within 4 weeks prior to day 1
* Cytochrome P450 CYP3A4 inducers and inhibitors within 4 weeks prior to day 1
* Intake of grapefruit, grapefruit juice, Seville oranges, or other products containing grapefruit or Seville oranges within 14 days prior to day 1
* UGT1A1 genotype of TA 7 in both alleles (homozygous UGT1A1*28) or TA 8 in either one or both alleles (hetero- or homozygous for UGT1A1*37)
* Major surgery within 4 weeks prior to day 1
* Undergone a liver or other organ transplant
* Concurrent treatment with other anti-cancer therapy
* Untreated central nervous system metastases
* Ongoing or active infection
* Chronic or acute GI disorders resulting in diarrhea
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of NKTR-102 and its metabolites | Day 1 through Day 42
  1 pre-dose PK measurements 14 post-dose PK measurements

SECONDARY OUTCOMES:
Safety and tolerability of NKTR-102 | Day 1 through Day 42
  Assessments are: physical examinations, vital signs, ECGs, AEs, and laboratory testing.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Gergel, MD, Study Director — Nektar Therapeutics
Locations (3):
- United States (3):
  - USC/LA County, Los Angeles, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - University Hospitals Case-Medical Center Seidman Cancer Center, Cleveland, Ohio